CLINICAL TRIAL: NCT01115569
Title: A Long-Term Open-Label Safety Study of Hydrocodone Bitartrate Controlled-Release Capsules With Flexible Dosing to Treat Subjects With Moderate to Severe Chronic Pain
Brief Title: Long-Term Study of Hydrocodone Bitartrate Controlled-release Capsules in Subjects With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX002-0802
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2014-03

CONDITIONS: Chronic Pain
Keywords: chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocodone Bitartrate (Experimental): Open-label, all patients fulfilling the protocol Inclusion/Exclusion criteria will receive HC-CR in a flexible dosing regimen.
  Interventions: Drug: Hydrocodone Bitartrate

INTERVENTIONS:
Drug: Hydrocodone Bitartrate — Open-Label, Capsule Strengths 10 mg, 20 mg, 30 mg, 40 mg, 50 mg; by mouth (PO) twice a day (BID) for up to 48 weeks
  Other Names: Hydrocodone Bitartrate Controlled Release (HC-CR)

SUMMARY:
This Phase 3, multi-center study will evaluate the long-term safety and tolerability of hydrocodone bitartrate controlled release capsule (HC-CR) at daily doses of 40 mg or more in subjects with moderate to severe chronic pain. Long-term maintenance of HC-CR efficacy will be evaluated.

DETAILED DESCRIPTION:
Subjects will go through screening, an open-label conversion and titration phase of up to 6 weeks followed by an open-label treatment phase for up to 48 weeks with a 2 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosed moderate to severe chronic pain condition treated with around-the-clock opioids for at least the past 3 months or in the Investigator's opinion qualify for around-the-clock opioid therapy for treatment of their pain
* Subjects must have been taking opioids at least 5 days/week for the past month at an average daily dose of at least 30 mg hydrocodone
* Subjects must be able to complete study procedures and attend clinic visits for 6 to 12 months
* Females subjects of childbearing potential must have a negative urine pregnancy test at the Screen Visit, and must consent to use a medically-acceptable method of contraception throughout the entire study period.
* Subjects must have had an adequate medical evaluation for the treatment of their underlying painful condition and appropriate primary medical/surgical therapies for the underlying condition
* Subjects must voluntarily provide written informed consent

Exclusion Criteria:

* Any clinically significant condition that would, in the opinion of the investigator, preclude study participation or interfere with the assessment of pain or increase the risk of opioid-related adverse events (AEs)
* A medical condition that, in the opinion of the Investigator, would compromise the subject's ability to swallow, absorb, metabolize, or excrete study drug
* A surgical procedure for pain within the last 3 months
* Uncontrolled blood pressure, i.e., a sitting systolic blood pressure >180 mm Hg or <90 mm Hg, and/or a sitting diastolic blood pressure >120 mm Hg or <50 mm Hg at Screening
* A body mass index (BMI) > 45 kg/m2
* A hospital anxiety and depression scale (HADS) score of >12 in either depression or anxiety subscales or an established history of any psychiatric disorder that is poorly controlled
* A clinically significant abnormality in clinical chemistry, hematology or urinalysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Gorgone, Study Director — Zogenix, Inc.
Locations (50):
- United States (50):
  - Arizona Research Center, Phoenix, Arizona
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Ortho Research, Little Rock, Arkansas
  - Pain Institute of California, Bakersfield, California
  - Providence Clinical Research, Burbank, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Scripps Clinic, Clinical Research, San Diego, California
  - Mountain View Clinical Research, Inc., Golden, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - National Pain Research Institute, Inc., Winter Park, Florida
  - Best Clinical Research, Decatur, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Better Health Clinical Research, Inc, Newnan, Georgia
  - Nautical Clinical Research, LLC, Boise, Idaho
  - Suburban Clinical Research, Bolingbrook, Illinois
  - International Clinical Research Institute, Inc., Leawood, Kansas
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Clinical Trials Managements, LLC, Mandeville, Louisiana
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - New England Center for Clinical Research, Internal Medicine and Cardiology Associates, LLC, Fall River, Massachusetts
  - Infinity Medical Research, Inc., North Dartmouth, Massachusetts
  - Mid-South Anesthesia Consultants, Southaven, Mississippi
  - Clinvest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Research West, LLC, Kalispell, Montana
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - New York University Pain Management Center, New York, New York
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Valley Medical Group, PC, Centerville, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Hometown Urgent Care and Research, Springfield, Ohio
  - Hillcrest Clinical Research, Inc., Oklahoma City, Oklahoma
  - Memorial Clinical Research DBA Angelique Barreto, MD, Oklahoma City, Oklahoma
  - Blair Medical Associates, Altoona, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - New England Center for Clinical Research, Inc., Cranston, Rhode Island
  - Renaissance Clinical Research and Hypertension Clinic, Dallas, Texas
  - The Clinical Research Center, LLC, Fort Worth, Texas
  - Heights Doctors Clinic, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Quality Research, Inc., San Antonio, Texas
  - West Side Medical, Clinton, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Advanced Pain Management, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 638 subjects treated with Hydrocodone Bitartate Extended Release (HC-ER) capsules in the Conversion/Titration Phase, 214 subjects discontinued early and 424 continued in the Maintenance HC-ER Treatment Phase; 285 subjects completed.
Groups:
- Open-label Hydrocodone Bitartrate Extended Release (HC-ER): Conversion/Titration Phase: HC-ER capsules daily for up to 6 weeks
- Open-label Hydrocodone Bitartrate Extended Release Capsules: Maintenance HC-ER Treatment Phase: Open-label, all patients fulfilling the protocol Inclusion/Exclusion criteria will receive HC-ER in a flexible dosing regimen.
  Hydrocodone Bitartrate: Open-Label, Capsule Strengths 10 mg, 20 mg, 30 mg, 40 mg, 50 mg; by mouth (PO) twice a day (BID) for up to 48 weeks
Period: Conversion/Titration Phase
Arm/Group | Open-label Hydrocodone Bitartrate Extended Release (HC-ER) | Open-label Hydrocodone Bitartrate Extended Release Capsules
Started | 638 | 0
Completed | 424 | 0
Not Completed | 214 | 0
Not completed — Adverse Event | 59 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 5 | 0
Not completed — Protocol Violation | 68 | 0
Not completed — Withdrawal by Subject | 26 | 0
Not completed — Non-Compliance with Study Drug | 53 | 0
Period: Maintenance Phase
Arm/Group | Open-label Hydrocodone Bitartrate Extended Release (HC-ER) | Open-label Hydrocodone Bitartrate Extended Release Capsules
Started | 0 | 424
Completed | 0 | 285
Not Completed | 0 | 139
Not completed — Adverse Event | 0 | 43
Not completed — Lost to Follow-up | 0 | 8
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 0 | 9
Not completed — Withdrawal by Subject | 0 | 27
Not completed — Non-Compliance with Study Drug | 0 | 48
Not completed — Administrative | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label Hydrocodone Bitartate Extended Release (HC-ER): Conversion/Titration Phase: HC-ER capsules daily for up to 6 weeks
Arm/Group | Open-label Hydrocodone Bitartate Extended Release (HC-ER)
Number analyzed (Participants) | 638
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 572
  >=65 years | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360
  Male | 278
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 107
  White | 518
  More than one race | 9
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 638

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Daily Pain
Description: Numeric Rating Scale (NRS) for Pain (0-10; where 0 = no pain, 10 = worst pain imaginable) recorded up to 54 weeks, starting at screening through end of study. Lower number equals better outcome.
Time Frame: 1 year
Population: The number of participants for analysis was determined by the safety population. Numeric Rating Scale (NRS) for Pain assessment was used. Measure is mean change in average daily pain intensity. Total number of participants providing end of study pain intensity score = 391.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Hydrocodone Bitartrate Extended Release Capsules: Maintenance HC-ER Treatment Phase: Open-label, all patients fulfilling the protocol Inclusion/Exclusion criteria will receive HC-CR in a flexible dosing regimen.
  Hydrocodone Bitartrate: Open-Label, Capsule Strengths 10 mg, 20 mg, 30 mg, 40 mg, 50 mg; by mouth (PO) twice a day (BID) for up to 48 weeks
Arm/Group | Open-label Hydrocodone Bitartrate Extended Release Capsules
Number analyzed (Participants) | 391
units on a scale | 0.921 (2.2)

2. Secondary Outcome: Maintenance of Efficacy
Description: Clinic Numeric Rating Scale (NRS), Brief Pain Inventory (BPI), Oswestry Disability Index, Hospital Anxiety and Depression Scale, Rescue Doses and Subject Global of Medication
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded up to 54 weeks, beginning at the Conversion and Titration Phase through 2 weeks after the last treatment administration (Treatment Phase).
Description: Subjects received a follow up phone call 14 days after the end of study to collect information regarding adverse events (AEs) or new serious AEs that occurred during this time period.
Groups:
- Conversion/Titration Phase: Conversion/Titration Phase: Hydrocodone Bitartrate Extended Release (HC-ER) capsules daily for up to 6 weeks
- Maintenance Treatment Phase: Maintenance Hydrocodone Bitartrate Extended Release (HC-ER) Treatment Phase: Open-label, all patients fulfilling the protocol Inclusion/Exclusion criteria will receive HC-CR in a flexible dosing regimen.
  Hydrocodone Bitartrate: Open-Label, Capsule Strengths 10 mg, 20 mg, 30 mg, 40 mg, 50 mg; by mouth (PO) twice a day (BID) for up to 48 weeks
Arm/Group | Conversion/Titration Phase | Maintenance Treatment Phase
Serious Adverse Events (participants affected / at risk) | 26/638 | 73/424
Other Adverse Events (participants affected / at risk) | 277/638 | 298/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion/Titration Phase (N=638) | Maintenance Treatment Phase (N=424)
Cystitis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrage (Gastrointestinal disorders) | 1 | 0
Osteoarthrtis (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blood potassium decreased (Investigations) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pathogen resistance (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intenstional overdose (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicidal attempt (Psychiatric disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conversion/Titration Phase (N=638) | Maintenance Treatment Phase (N=424)
Constipation (Gastrointestinal disorders) | 72 | 53
Nausea (Gastrointestinal disorders) | 68 | 42
Somnolence (Nervous system disorders) | 49 | 18
Headache (Nervous system disorders) | 48 | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 47
Vomiting (Gastrointestinal disorders) | 26 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 33
Urinary tract infection (Infections and infestations) | 6 | 28
Fall (Injury, poisoning and procedural complications) | 8 | 25
Upper respiratory tract infection (Infections and infestations) | 7 | 25
Nasopharyngitis (Infections and infestations) | 11 | 24
Anxiety (Psychiatric disorders) | 8 | 23
Sinusitis (Infections and infestations) | 9 | 23
Insomnia (Psychiatric disorders) | 24 | 21
Fatigue (General disorders) | 23 | 15
Diarrhoea (Gastrointestinal disorders) | 20 | 17
Dizziness (Nervous system disorders) | 18 | 13
Oedema peripheral (General disorders) | 14 | 14
Pruritus allergic (Skin and subcutaneous tissue disorders) | 13 | 0
Bronchitis (Infections and infestations) | 10 | 20
Influenza (Infections and infestations) | 4 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 18
Depression (Psychiatric disorders) | 6 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 16
Pyrexia (General disorders) | 11 | 15
Contusion (Injury, poisoning and procedural complications) | 4 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14
Muscle strain (Injury, poisoning and procedural complications) | 9 | 13
Migraine (Nervous system disorders) | 5 | 11
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 11
Gastroenteritis viral (Infections and infestations) | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Paraesthesia (Nervous system disorders) | 1 | 9
Pneumonia (Infections and infestations) | 3 | 9
Toothache (Gastrointestinal disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days